CLINICAL TRIAL: NCT05916456
Title: Investigation of the Validity and Reliability of the Hand10 Questionnaire in Individuals With Carpal Tunnel Syndrome
Brief Title: Hand10 Questionnaire in Individuals With Carpal Tunnel Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Neslihan Torun, MSc, Hasan Kalyoncu University
Other Study IDs: HasanKU''
Record Dates: First submitted 2023-06-07; First posted 2023-06-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; DASH questionnaire; Boston carpal tunnel syndrome questionnaire; HAND10 questionnaire; validity and reliability
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Hand10 Questionnaire — The Hand10 Questionnaire is a questionnaire consisting of 10 short questions used in the evaluation of upper extremity diseases. These questions are easy to understand and illustrated questions. Unlike other questionnaires, thanks to these features, it can be used in adults as well as in the elderly and children. Tore et al. In their study, the internal consistency of Hand10 was evaluated with Cronbach's alpha value according to statistical results and found it to be 0.919. According to these results, it has been determined that Hand10 is a reliable and valid assessment tool for patients with upper extremity disorders in the Turkish population.
Diagnostic Test: DASH Questionnaire — DASH Questionnaire is one of the widely used questionnaires consisting of 30 items. There are five options for each answer. While getting answers ranging from 1 to 5; 1 means no symptoms and 5 means very severe symptoms. The total DASH score ranges from 0 to 100; 0 means no injury and 100 means serious injury. Contrary to the Hand10 questionnaire, DASH was not suitable for assessing upper extremity disorders in patients over 65 years of age.
Diagnostic Test: Boston carpal tunnel syndrome questionnaire — Boston carpal tunnel syndrome questionnaire (BKTSA) will be used to evaluate the functionality level and symptom severity of the patients. In this questionnaire, which consists of 2 parts: symptom severity and functional capacity, the average score for each part will be calculated by dividing the total score obtained by the number of questions. An increased score indicates decreased functional capacity and increased symptom severity.

SUMMARY:
Hand10 questionnaire, Boston Carpal Tunnel Syndrome Questionnaire and Arm Shoulder Questionnaire for patients with carpal tunnel syndrome and Hand Deficiencies Questionnaire (DASH) will be applied one week apart to investigate the validity of the questionnaire.

Test-retest reliability and internal consistency will be determined using Intraclass Correlation Coefficient analysis and Cronbach alpha, respectively. The validity of Hand10 in individuals with CST will be determined using the Pearson Correlation Coefficient analysis, the Arm, Shoulder, and Hand Disability Questionnaire and the Boston Carpal Tunnel Syndrome Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteer for treatment
* 18-70 years old patients
* With patients diagnosed with CTS

Exclusion Criteria:

-Patients who have had surgery on the wrist area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study will be conducted with individuals between the ages of 18-70 who have been diagnosed with CTS.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The validity and reliability of the Hand10 questionnaire to individuals with carpal tunnel scan included | 3 month
  Patients diagnosed with Carpal tunnel by the doctor

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Universty, Gaziantep, Sahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No